CLINICAL TRIAL: NCT04469543
Title: A Retrospective Cohort Study: Influence of MTHFR C677T and A1298C Polymorphisms on the Survival of Pediatric Patients With Non-Hodgkin's Lymphoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiao-Fei Sun, MD, Sun Yat-sen University
Other Study IDs: SCCCG-NHL2017
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Pediatric Non-Hodgkin Lymphoma
Keywords: MTHFR C677T polymorphism；A1298C; Pediatric Non-Hodgkin Lymphoma；Survival.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- MTHFR polymorphism

SUMMARY:
The primary purpose of this retrospective study was to investigate the influence of methylenetetrahydrofolate reductase (MTHFR) C677T/A1298C polymorphism on the survival of pediatric patients with Non-Hodgkin lymphoma (NHL) treated with modified NHL-BFM95 protocol in south China.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≤ 18 years;
2. newly diagnosed as the four main categories of NHL(Burkitt's lymphoma, lymphoblastic lymphoma, anaplastic large cell lymphoma, and diffuse large B-cell lymphoma) between 2014 and 2020;
3. treated according to the modified BFM95 protocol.

Exclusion Criteria:

1. aged > 18 years;
2. not newly diagnosed as the four main categories of NHL between 2014 and 2020;
3. treated according to chemotherapeutic regimens except for the modified BFM95 protocol.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We reviewed all the medical records of the patients who met the inclusion criteria in Sun Yat-sen University Cancer Center
Sampling Method: Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Death | About six years
  Overall survival time was calculated from the time of initial diagnosis to death
Events including progression, relapse, and secondary cancer | About six years
  Event-free survival (EFS) time was calculated from the time of initial diagnosis to first event.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided